CLINICAL TRIAL: NCT00093990
Title: A Randomized Study of Tipifarnib Versus Best Supportive Care (Including Hydroxyurea) in the Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML) in Subjects 70 Years or Older (Farnesyl Transferase Inhibition Global Human Trials AML 301 [F.I.G.H.T. AML 301])
Brief Title: Tipifarnib Versus Best Supportive Care in the Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004372
Record Dates: First submitted 2004-10-07; First posted 2004-10-11 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Myeloid leukemia acute disease; Tipifarnib; Bone marrow aspirate
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tipifarnib

INTERVENTIONS:
Drug: Tipifarnib;Zarnestra; R115777

SUMMARY:
The purpose of this study is to determine the effectiveness of tipifarnib in patients aged 70 or more with acute myeloid leukemia. Tipifarnib belongs to a class of drugs called Farnesyl Transferase Inhibitors (FTI). It blocks proteins that make leukemia cells grow.

DETAILED DESCRIPTION:
This study tests the safety and effectiveness of the experimental drug, tipifarnib in older patients who have acute myeloid leukemia (AML). The purpose of this study is to test if tipifarnib can make patients with leukemia live longer. In this study, half the patients will receive tipifarnib and half of the patients will receive the standard treatment. The standard treatment will help to control the symptoms of AML and may include hydroxyurea to lower levels of circulating leukemia cells. Tipifarnib or the standard treatment will be given until the patient's leukemia gets better, or until they experience unacceptable side effects, or until the patient or study doctor decide to stop the study medication. Patients assigned to tipifarnib will be given tipifarnib tablets. Patients should take 6 tablets with food in the morning and 6 tablets with food in the evening, for 21 days in a row. Patients will not take tipifarnib for the next 7 days. This 28 day period is called a cycle. The rest period may be extended beyond 7 days depending on how well the patients tolerate the treatment. Patients will return to the study clinic every week and to visit their study doctor at least every two weeks. A blood draw for routine tests will be done every week. Depending on how your disease is doing, a bone marrow aspiration may be done at the end of every cycle. When patients finish treatment with the study medication, or if they leave the study early, they will be asked to see your doctor for one last visit. Routine laboratory tests will be done. After this visit the study doctor will continue to check with patients to see how they are doing and if they have started a new treatment for leukemia. This check will be made every 30 days and may be made by phone to the patient or to their health care provider. Tipifarnib; six 100 mg in a film coated, compressed tablets are given orally twice a day at for 21 consecutive days on a 28-day cycle schedule.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or re-lapsing AML
* Patient not medically fit for combination induction chemotherapy
* Pathologic confirmation of AML (= or > 20% bone marrow leukemic blasts)
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.

Exclusion Criteria:

* Previous cytotoxic or biologic treatment for AML
* Acute promyelocytic leukemia (APL)
* Central nervous system leukemia
* Uncontrolled systemic infection
* Uncompensated disseminated intravascular coagulation
* Symptomatic neuropathy of grade 2 or worse
* Known allergy to imidazole drugs.

Ages: 70 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 457 (Actual)
Dates: Start 2004-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Compare patients treated with tipifarnib and patients treated with best supportive care: progression-free survival; complete remission rate; rate of morphologic leukemia-free state; one-year survival estimate and health resources utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Harousseau JL, Martinelli G, Jedrzejczak WW, Brandwein JM, Bordessoule D, Masszi T, Ossenkoppele GJ, Alexeeva JA, Beutel G, Maertens J, Vidriales MB, Dombret H, Thomas X, Burnett AK, Robak T, Khuageva NK, Golenkov AK, Tothova E, Mollgard L, Park YC, Bessems A, De Porre P, Howes AJ; FIGHT-AML-301 Investigators. A randomized phase 3 study of tipifarnib compared with best supportive care, including hydroxyurea, in the treatment of newly diagnosed acute myeloid leukemia in patients 70 years or older. Blood. 2009 Aug 6;114(6):1166-73. doi: 10.1182/blood-2009-01-198093. Epub 2009 May 21. PMID 19470696